CLINICAL TRIAL: NCT00255177
Title: A Randomized, Open-label Phase II Trial of the Anti-HCV Activity and Safety of VGX-410 (Mifepristone) at 3 Dose Levels in HCV Infected Patients
Brief Title: Antiviral Activity and Safety of 3 Different Doses of Mifepristone in Hepatitis C Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VGX Pharmaceuticals, LLC (Industry)
Responsible Party: VGX Pharmaceuticals, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VT003; Viral Genomix, Inc. (VGX); 450 Sentry Parkway; Blue Bell, PA 19422; C. Jo White, M.D.
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-10

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 150 mg daily (Active Comparator)
  Interventions: Drug: VGX-410 (Mifepristone)
- 300mg daily (Active Comparator)
  Interventions: Drug: VGX-410 (Mifepristone)
- 300mg twice daily (Active Comparator)
  Interventions: Drug: VGX-410 (Mifepristone)

INTERVENTIONS:
Drug: VGX-410 (Mifepristone) — VGX-410 tablets taken daily or twice daily for 28 days
  Other Names: Mifepristone
  Arms: 150 mg daily; 300mg daily; 300mg twice daily
Drug: Placebo — Placebo for VGX-410 tablets taken daily or twice daily for 28 days
  Arms: Placebo

SUMMARY:
Hepatitis C virus (HCV) infects approximately 170 million people worldwide. The current standard- of- care therapy of chronic HCV infection is a regimen of subcutaneously administered (pegylated)-interferon-α and ribavirin for 24 weeks (for genotypes 2 and 3) to 48 weeks (for genotype 1). The sustained viral response rates (SVR) in patients infected with genotypes 2 and 3 are ~80% but remain <50% in patients infected with genotype 1. The treatment is quite toxic with approximately 30% of patients experiencing adverse events (i.e. depression, fever, anemia, fatigue) requiring dose reduction or discontinuation of therapy. This regimen is contraindicated in women who are pregnant and in patients with decompensated liver disease. The absence of acceptable therapies for many patients with HCV infections makes new therapies desirable for this disease.

DETAILED DESCRIPTION:
The 341-nucleotide 5' non-translated region is the most conserved part of the hepatitis C virus (HCV) genome. It contains a highly structured internal ribosomal entry site (IRES) that mediates cap-independent initiation of translation of the viral polyprotein by a mechanism that is unprecedented in eukaryotes. The first step in translation initiation is assembly of eukaryotic initiation factor (eIF) 3, eIF2, GTP, initiator tRNA and a 40S ribosomal subunit into a 43S preinitiation complex (1, 2). The IRES contains sites that bind independently with the eIF3 and 40S ribosomal subunit components of 43S complexes, and structural determinants that ensure the correct spatial orientation of these binding sites so that the 48S complex assembles precisely at the initiation codon. Since inhibiting this early translation of viral protein should block HCV replication downstream, this early critical step in replication is of great interest as a drug target. All genotypes of HCV use the same pathway; this drug target should be effective for all HCV genotypes.

VGX-410 represents the first drug in a novel class of HCV IRES inhibitors under development. VGX-410 is an orally active and bioavailable, small-molecule, organic drug. Because a related formulation of mifepristone has been previously approved by the FDA for another indication (medical abortion), there are pre-existing data from animal toxicity tests showing the safety of this compound at very high doses (5 mg/kg for 6 months in rats and macaques). In addition, chronic administration (up to 200 mg/day) of this compound for the experimental treatment of a variety of malignant and non-malignant conditions has been well tolerated in non-HCV-infected subjects for up to 1 year (3-6).

In cell culture tests, VGX-410 has been shown to be effective in inhibiting HCV replication with the 50% and 90% effective antiviral concentrations (EC50 and EC90) of 2 and 10 μM, respectively. Furthermore, VGX-410 was shown to act synergistically with interferon-a (IFN-a), the most widely-used drug treatment option available today. When used in combination with a low dose IFN-a at 1 IU/ml, EC90 of VGX-410 was reduced to 3 µM. Moreover, since VGX-410 inhibits viral replication by blocking the cellular protein complex for HCV IRES, there is reduced potential for viral mutation and resistance to this drug.

From these in vitro data, we would expect to observe 50 to 90% anti-HCV effects in humans at serum drug concentrations of 2 to 10 μM, respectively. Moreover, we compiled the drug concentration results from several previously-reported clinical data on the level of steady-state concentrations in patients who took repeat daily doses of mifepristone (>4 days). For instance, repeated oral administration of 100 and 200-mg mifepristone daily for 4 days achieved maximum plasma levels of 4.5 and 5.4 μM, respectively (9).

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C infection for ≥ 1 year. Viral load at entry will be measured by the Amplicor Hepatitis C Virus Test Version 2.0 (Roche Molecular Systems; Plesasanton, CA) and genotyped by Trugene HCV 5'NC Genotyping kit (Visible Genetics; Toronto, Canada) performed within 90 days prior to study entry by a lab(s) certified for the assays.
* Male or female ages 18-65 years, inclusive.
* Plasma hepatitis C RNA of >105 copies/mL (or equivalent international units)
* Laboratory values: stable hepatic, renal, and hematological indices obtained within 30 days prior to study entry, as follows:

  * Absolute neutrophil count (ANC) >= 750/mm³
  * Hemoglobin >= 10.0 g/dL
  * Platelet count >= 100,000/mm3
  * Creatinine <= 2 x ULN
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase <= 3 x ULN
  * Total bilirubin <= 3 x ULN
  * Albumin >= 3 g/dL
  * Normal PT and PTT
  * Serum lipase <= 1.5 x ULN
  * TSH within normal limits (0.5-6.0 mIU/L)
  * Morning plasma cortisol >= 20 µg/dL
  * Normal fasting glucose
  * Urinalysis free of clinically significant abnormalities NOTE: Fasting is defined as no oral intake except water for at least 8 hours prior to the study visit.
* Female subjects of reproductive potential (girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months or have not undergone surgical sterilization [e.g., hysterectomy, bilateral oophorectomy, or salpingotomy]) must have a negative spot urine pregnancy test result (with a sensitivity of at least 50 mIU/mL) performed at entry, before initiating study medication.
* All subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, donate sperm, or in vitro fertilization). If participating in sexual activity that could lead to pregnancy, the subject/partner must agree to use two reliable methods of contraception simultaneously (condoms with a spermicidal agent; or a diaphragm or cervical cap with spermicide) while on study drug and for 30 days after stopping the medication.
* Female subjects, who are not of reproductive potential, are eligible without requiring the use of contraception. Male subjects must use a condom with every sexual act that could lead to pregnancy.

NOTE: Acceptable documentation of sterilization is either written or oral documentation communicated by clinician or clinician's staff of one of the following: physician report/letter: operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy); discharge summary; laboratory report of azoospermia; or FSH measurement elevated into the menopausal range as established by the reporting laboratory.

* Karnofsky performance score >= 80 within 30 days prior to study entry.
* Ability and willingness of subject to give written informed consent.
* Willingness to return for a follow-up visit on day 56.
* Subjects taking any precautionary concomitant medications (see section 5.2.2) must be on stable doses for >8 weeks prior to study entry and have no plans to change medications or doses for the duration of the study.

Exclusion Criteria:

* Receipt of anti-hepatitis C therapy within the 4 weeks prior to study entry or intent to initiate ant-hepatitis C therapy within 60 days after entry.
* Clinical evidence of cirrhosis or decompensated liver failure.
* Chronic or acute adrenal failure, history of active hepatitis B, HIV-1 infection, porphyrias, known moderate to severe cirrhosis, hemorrhagic disorders, concurrent anticoagulant therapy, any prior pituitary tumor, surgery, radiation treatment, or pituitary failure.
* Diabetes requiring treatment with oral hypoglycemics or insulin therapy.
* Pregnancy within 90 days prior to study entry.
* Breast-feeding.
* Dysfunctional uterine bleeding within the 12 months prior to study entry.
* Any current hormonal contraception or IUD use.
* Use of drugs that are inhibitors or inducers of metabolism by the CYP 3A4 within 7 days of study entry.
* Use of systemic corticosteroids or hormonal agents within 90 days prior to study entry.
* Use of any cytotoxic chemotherapy, immunomodulators or investigational therapy within 90 days prior to study entry.
* Any vaccination within 30 days prior to study entry.
* Allergy to mifepristone or its formulation.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirement.
* Weight < 40 kg.
* Any other condition thought by the investigator that may interfere with the patient's ability to comply with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Bacon, M.D., Principal Investigator — St. Louis University; Pablo Tebas, M.D., Principal Investigator — University of Pennsylvania; George Wu, MD, Principal Investigator — University of Connecticut; Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center
Locations (4):
- United States (4):
  - University of Connecticut, Farmington, Connecticut
  - Orlando Clinical Research Center, Orlando, Florida
  - Saint Louis University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Kieft JS, Zhou K, Jubin R, Doudna JA. Mechanism of ribosome recruitment by hepatitis C IRES RNA. RNA. 2001 Feb;7(2):194-206. doi: 10.1017/s1355838201001790. PMID 11233977

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | VGX-410 150mg Daily | VGX-410 300mg Daily | VGX-410 300mg Twice Daily
Started | 11 | 14 | 13 | 6
Completed | 9 | 13 | 12 | 4
Not Completed | 2 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VGX-410 150mg Daily | VGX-410 300mg Daily | VGX-410 300mg Twice Daily | Total
Number analyzed (Participants) | 11 | 14 | 13 | 6 | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 48.0 (6.9) | 45.4 (6.9) | 47.4 (9.2) | 52.0 (3.7) | 47.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 2 | 14
  Male | 6 | 10 | 10 | 4 | 30
Region of Enrollment [Number; unit: participants]
  United States | 11 | 14 | 13 | 6 | 44

OUTCOME MEASURES:

1. Primary Outcome: Mean Log Change in Viral Load From Baseline (Day 1) to Day 28
Description: Mean log change in HCV RNA viral load (significant reduction is considered >0.5 log 10) from baseline (Day 1) following once or twice daily dosing for 28 days at the 28 day timepoint
Time Frame: Baseline (Day 1) to Day 28
Measure: Log Mean (Standard Deviation); unit: copies/mL on log scale
Arm/Group | Placebo | VGX-410 150mg Daily | VGX-410 300mg Daily | VGX-410 300mg Twice Daily
Number analyzed (Participants) | 9 | 14 | 11 | 6
copies/mL on log scale | 0.30 (0.45) | 0.00 (0.30) | 0.18 (0.32) | 0.04 (0.39)

ADVERSE EVENTS:
Time Frame: AEs that occurred during treatment period (Days 1-28)
Arm/Group | Placebo | VGX-410 150mg Daily | VGX-410 300mg Daily | VGX-410 300mg Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14 | 1/13 | 0/6
Other Adverse Events (participants affected / at risk) | 11/11 | 14/14 | 13/13 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=11) | VGX-410 150mg Daily (N=14) | VGX-410 300mg Daily (N=13) | VGX-410 300mg Twice Daily (N=6)
Generalized Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0/11 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | VGX-410 150mg Daily (N=14) | VGX-410 300mg Daily (N=13) | VGX-410 300mg Twice Daily (N=6)
Ear and Labyrinth Disorders (Ear and labyrinth disorders) | 0 (0) | 1 | 0 (0) | 0 (0)
Eye Disorders (Eye disorders) | 0 (0) | 1 | 3 | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 | 2 | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 (0) | 4 | 5 | 2
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 | 1 | 1
Fatigue (General disorders) | 3 | 6 | 3 | 1
Oedema Peripheral (General disorders) | 0 (0) | 2 | 2 | 0 (0)
Immune System Disorders (Immune system disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
Infections and Infestations (Infections and infestations) | 2 | 0 (0) | 1 | 0 (0)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 0 (0) | 2 | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 8 | 8 | 9 | 4
Aspartate Aminotransferase Increased (Investigations) | 6 | 8 | 9 | 5
Blood Albumin Abnormal (Investigations) | 1 | 1 | 2 | 1
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 | 1 | 2
Blood Cholesterol Abnormal (Investigations) | 1 | 3 | 1 | 1
Blood Glucose Abnormal (Investigations) | 7 | 8 | 8 | 4
Blood Glucose Increased (Investigations) | 1 | 1 | 0 (0) | 1
Blood Potassium Increased (Investigations) | 1 | 1 | 0 | 1
Blood Triglycerides Abnormal (Investigations) | 1 | 2 | 0 | 0
Haemoglobin Decreased (Investigations) | 2 | 2 | 2 | 0
Neutrophil Count Decreased (Investigations) | 2 | 2 | 2 | 1
Platelet Count Decreased (Investigations) | 1 | 1 | 3 | 1
White Blood Cell Count Decreased (Investigations) | 2 | 2 | 0 | 2
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 3 | 0
Dizziness Postural (Nervous system disorders) | 1 | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 5 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 0 | 3 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1
Surgical and Medical Procedures (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hot Flush (Vascular disorders) | 1 | 3 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No